CLINICAL TRIAL: NCT02816281
Title: Scheduled Elective Surgical Case Cancellation in Siriraj Hospital, a Thai University Hospital: Evaluation and Identification of the Reasons
Brief Title: Scheduled Elective Surgical Case Cancellation in Siriraj: Evaluation and Identification of the Reasons
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mingkwan Wongyingsinn, MD, Assistant Professor, Siriraj Hospital
Other Study IDs: SIRB305
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Peer Review, Research
Keywords: Surgical case cancellation; Pre-operative assessment clinic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Reasons of case cancellation: will be recorded and categorized into 6 groups including
  1. patient issue such as surgery refusal, no show on the day of surgery, transport problems
  2. facility such as equipment needs, improper estimate case time, case bumps
  3. Surgeon unavailable, due to administrative schedules and other problems or changed line of management respectively
  4. anesthesiologist fail to adequately prepare the patient, lead to some misunderstanding communication such as NPO violation, preoperative drug error
  5. medical condition that may impact the patient's ability to endure anesthesia techniques or surgical procedure
  6. miscellaneous.

SUMMARY:
A retrospective cross-sectional analytic study to evaluation and identification of the reasons about Scheduled elective surgical case cancellation in Siriraj Hospital, reason of cancellation will be extracted from hospital medical record of each case, reviewed and divided into 2 groups, with SiPAC and without SiPAC consultation. Primary outcomes are the incidence of cancelled case and causes of the cancellation and secondary outcome that will be identified for areas of improvement.

DETAILED DESCRIPTION:
After approval by the Siriraj Institutional Review Board. All data of case cancellation on scheduled elective surgical procedures will be retrieved from database of the department of Anesthesiology, Faculty of Medicine Siriraj Hospital. Then, reason of cancellation will be extracted from hospital medical record of each case. All cases will be checked in database of SiPAC, department of Anesthesiology, Faculty of Medicine Siriraj Hospital to confirm whether each patient was preoperatively consulted. All patients having cancellation on scheduled elective surgery in the period of one year will be reviewed. Exclusion criteria is 1) patients having emergency or urgency surgery which means patients' names were not appeared in the surgical schedules 2) having missing key medical information.

Admission records and patient charts will be reviewed and divided into 2 groups, with SiPAC and without SiPAC consultation. Primary outcomes are the incidence of cancelled case and causes of the cancellation which will be recorded and categorized into 6 groups including 1) patient issue such as surgery refusal, no show on the day of surgery, transport problems 2) facility such as equipment needs, improper estimate case time, case bumps 3) Surgeon unavailable, due to administrative schedules and other problems or changed line of management respectively 4) anesthesiologist fail to adequately prepare the patient, lead to some misunderstanding communication such as NPO violation, preoperative drug error 5) medical condition that may impact the patient's ability to endure anesthesia techniques or surgical procedure 6) miscellaneous. The results compared between in patients with and without SiPAC consultation will be analyzed as a secondary outcome that will be identified for areas of improvement.

ELIGIBILITY:
Inclusion Criteria:

* all data of case cancellation on scheduled elective surgical procedures

Exclusion Criteria:

* patients having emergency or urgency surgery which means patients' names were not appeared in the surgical schedules

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All data of case cancellation on scheduled elective surgical procedures will be retrieved from database of the department of Anesthesiology, Faculty of Medicine Siriraj Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2760 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Reasons of case cancellation | 1 year
  all caused of the cancellation will be recorded and categorized into 6 groups

SECONDARY OUTCOMES:
Incidence of case cancellation | 1 year
  Incidence of case cancellation

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, MD, MSc, Principal Investigator — Faculty of Medicine Siririaj Hospital
Locations (1):
- Siriraj hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vongchaiudomchoke W, Wongcharoen P, Wongyingsinn M. The impact of a preanesthesia assessment clinic on scheduled elective case cancelations at a Thai university hospital. Medicine (Baltimore). 2023 Aug 25;102(34):e34823. doi: 10.1097/MD.0000000000034823. PMID 37653830